CLINICAL TRIAL: NCT05838001
Title: Efficacy and Accuracy of Combined Localization Versus Single Localization in Non-palpable Breast Cancer After Neo-adjuvant Therapy : a Prospective Randomized Control Trial.
Brief Title: Efficacy and Accuracy of Combined Localization Versus Single Localization in Non-palpable Breast Cancer After Neoadjuvant Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chang Gong, Clinical Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-129-02
Record Dates: First submitted 2023-04-02; First posted 2023-05-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Breast-conserving Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients after neoadjuvant therapy-combined localization (Experimental)
  Interventions: Procedure: Wire-guided localization and marker clip localization
- patients after neoadjuvant therapy-single localization (Active Comparator)
  Interventions: Procedure: marker clip localization

INTERVENTIONS:
Procedure: Wire-guided localization and marker clip localization — Positioning guide wire and marker clip in the center of the breast lesion
  Arms: patients after neoadjuvant therapy-combined localization
Procedure: marker clip localization — Positioning marker clip in the center of the breast lesion
  Arms: patients after neoadjuvant therapy-single localization

SUMMARY:
The standard method for localizing non-palpable breast cancer is currently clip localization, its positive margin rate still remains around 20-50%. This study aims to compare the accuracy and efficacy of single vs. combined breast tissue markers in localizing non-palpable breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. female patients, age≥18 year
2. A score of ≥ 2 on the Eastern Cooperative Oncology Group scale
3. Patients pathologically diagnosed with breast cancer by core-needle biopsy, received neoadjuvant treatment and the lesion becomes non-palpable before enrollment.
4. Patients are willing to undergo breast conserving surgery and have no contraindications to breast conserving surgery

Exclusion Criteria:

1. Inflammatory breast cancer or Paget's disease
2. Breast deformities and other conditions that impact breast conservation success rate
3. Patients with contraindications to breast-conserving surgery, as well as those with systemic diseases, mental disorders, or other subjective reasons that may affect their ability to participate in the trial. Patients with severe bleeding disorders or coagulation disorders were also excluded.
4. Pregnancy or lactation
5. Patients with hook-wire, radioactive 125I seed or other localization techniques in the breast cancer lesions before enrollment
6. Patients with stage IV diseases or unresectable lesions in either breast
7. Patients combined with other diseases that may affect survival
8. Patients with multicentric breast cancer lesions or lesions > 5 cm in diameter on imaging examinations
9. Patients who have previously undergone radical mastectomy for ipsilateral breast cancer or chest wall radiotherapy
10. Patients with history of ipsilateral breast cancer radical mastectomy or chest wall radiotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Marginal positive rate | up to 3 months
  Proportion of patients with positive margin (intraoperative freezing and postoperative pathological margin tissue showing cancer)

SECONDARY OUTCOMES:
Re-operation rate. | up to 3 months
  the proportion of patients which have a positive margin and requires a re-operation
The proportion of breast-conserving surgery. | up to 3 months
  It refers to the proportion of patients who have successfully undergone breast-conserving surgery.
IDFS | 2 years, 3 years, and 5 years
  Time from surgery to the first occurrence of local, distant disease recurrence, or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China